CLINICAL TRIAL: NCT06608056
Title: Comparing Opioid Vs Non Opioid Analgesics for Postoperative Pain Management in Unilateral Primary Open Inguinal Hernia Repair
Brief Title: Comparing Opioids Vs NSAIDs for Postoperative Pain Management in Unilateral Primary Open Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Air Force (PAF) Hospital Islamabad (Other)
Responsible Party: Principal Investigator, Syed Moiz Ahmed, Post-graduate resident, Principle Investigator, Department of General Surgery, Pakistan Air Force (PAF) Hospital Islamabad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SGR-2021-137-2499-2; SGR-2021-137-2499-2 (Other: PAF Hospital ethical committee)
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Inguinal Hernia Unilateral; Pain Management
Keywords: Lichtenstein repair; ketorolac; tramadol; opioid; visual analogue score; non-steroidal anti-inflammatory drugs
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tramadol (Experimental): Patients received injection tramadol 50 mg intravenously every 8 hourly following surgery
  Interventions: Drug: Pain management after surgery
- Ketorolac (Experimental): Patients received injection tramadol 30 mg intravenously every 8 hourly following surgery
  Interventions: Drug: Pain management after surgery

INTERVENTIONS:
Drug: Pain management after surgery — Patients in Group A received injection tramadol 50mg intravenously every 8 hours following surgery. Patients in Group B received injection ketorolac 30mg intravenously every 8 hours following surgery.

SUMMARY:
To control post-operative pain, multiple drugs are available, and in the western countries opioids are preferred. However, they have their own side effects, and so to reduce their dependence, multiple adjuncts are used. We compared the use of opioids vs just non steroidal anti-inflammatory drugs on post-operative pain control following inguinal hernia surgery

DETAILED DESCRIPTION:
Inguinal hernia repair is one of the most common surgeries performed by general surgeons worldwide. The preferred procedure for primary open inguinal hernias is open mesh repair (tension-free)-also called Lichtenstein repair. Opioids remain the mainstay for post-operative analgesia, however, they have a tendency for dependence along with other side effects. Non-steroidal anti-inflammatory drugs (NSIADs) have been used as adjuncts to decrease the use of opioids, however, usually NSAIDs are not used in isolation following surgery. We compared post-operative analgesia following primary open inguinal hernia repair, with patients receiving only opioids vs patients only receiving NSAIDs. 60 patients were randomized in to 2 groups. Group A patients received tramadol injection (opioid) every 8 hours, while patients in Group B received injection ketorolac (NSAID) every 8 hourly. Pain was measured using visual analogue score at 2-, 6-, 12- and 24-hours following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective primary unilateral open inguinal hernia repair under spinal anesthesia - Lichtenstein repair with prolene mesh
* ASA I or II
* Ages 18 - 65

Exclusion Criteria:

* Patient on chronic pain meds
* Patient receiving analgesics 24hrs prior to surgery
* Incarcerated or strangulated hernia or recurrent hernia
* BMI >40
* Allergic to medications being tested in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale - pain score | 2-, 6-, 12-, 24-hours following surgery
  Visual analogue score to quantify pain following laparoscopic cholecystectomy. Maximum value is 10 (which means worst pain), and minimum value is 0 (which means no pain).

SECONDARY OUTCOMES:
Flatus | within 24 hours following surgery
  Time to passing flatus
nausea/vomiting | within 24 hours following surgery
  time when nausea/vomiting was not present in the patient
Time to ambulation | within 24 hours following surgery
  time after surgery when the patient started ambulating
rescue analgesia | within 24 hours following surgery
  number of times rescue analgesia was used
Mean arterial pressure | 2-, 6-, 12-, 24-hours following surgery
  systolic and diastolic blood pressures were measured for the patients at intervals, and then mean arterial pressures were calculated
Heart rate | 2-, 6-, 12-, 24 hours
  Heart rate was measured at intervals in beats per minute
oxygen saturation | 2-, 6-, 12-, 24 hours
  oxygen saturation was noted at intervals

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan Air Force Hospital, Islamabad, Capital Territory, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bugada D, Lavand'homme P, Ambrosoli AL, Klersy C, Braschi A, Fanelli G, Saccani Jotti GM, Allegri M; SIMPAR group. Effect of postoperative analgesia on acute and persistent postherniotomy pain: a randomized study. J Clin Anesth. 2015 Dec;27(8):658-64. doi: 10.1016/j.jclinane.2015.06.008. Epub 2015 Aug 30. PMID 26329661
- [Background] Zende, A.M. and R.R. Bhosale, Comparison of postoperative analgesic efficacy and safety of parecoxib and ketorolac in patients of inguinal hernia. International Journal of Basic and Clinical Pharmacology, 2013. 2(4): p. 414-20.
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] De Oliveira GS Jr, Agarwal D, Benzon HT. Perioperative single dose ketorolac to prevent postoperative pain: a meta-analysis of randomized trials. Anesth Analg. 2012 Feb;114(2):424-33. doi: 10.1213/ANE.0b013e3182334d68. Epub 2011 Sep 29. PMID 21965355
- [Background] Pavy TJ, Paech MJ, Evans SF. The effect of intravenous ketorolac on opioid requirement and pain after cesarean delivery. Anesth Analg. 2001 Apr;92(4):1010-4. doi: 10.1097/00000539-200104000-00038. PMID 11273941
- [Background] Chen JY, Wu GJ, Mok MS, Chou YH, Sun WZ, Chen PL, Chan WS, Yien HW, Wen YR. Effect of adding ketorolac to intravenous morphine patient-controlled analgesia on bowel function in colorectal surgery patients--a prospective, randomized, double-blind study. Acta Anaesthesiol Scand. 2005 Apr;49(4):546-51. doi: 10.1111/j.1399-6576.2005.00674.x. PMID 15777304
- [Background] National Academies of Sciences, Engineering, and Medicine; Health and Medicine Division; Board on Health Sciences Policy; Committee on Pain Management and Regulatory Strategies to Address Prescription Opioid Abuse; Phillips JK, Ford MA, Bonnie RJ, editors. Pain Management and the Opioid Epidemic: Balancing Societal and Individual Benefits and Risks of Prescription Opioid Use. Washington (DC): National Academies Press (US); 2017 Jul 13. Available from http://www.ncbi.nlm.nih.gov/books/NBK458660/ PMID 29023083
- [Background] Goettsch WG, Sukel MP, van der Peet DL, van Riemsdijk MM, Herings RM. In-hospital use of opioids increases rate of coded postoperative paralytic ileus. Pharmacoepidemiol Drug Saf. 2007 Jun;16(6):668-74. doi: 10.1002/pds.1338. PMID 17072916
- [Background] Barletta JF, Asgeirsson T, Senagore AJ. Influence of intravenous opioid dose on postoperative ileus. Ann Pharmacother. 2011 Jul;45(7-8):916-23. doi: 10.1345/aph.1Q041. Epub 2011 Jul 5. PMID 21730280
- [Background] Garimella V, Cellini C. Postoperative pain control. Clin Colon Rectal Surg. 2013 Sep;26(3):191-6. doi: 10.1055/s-0033-1351138. PMID 24436674
- [Background] Kehlet H, Holte K. Effect of postoperative analgesia on surgical outcome. Br J Anaesth. 2001 Jul;87(1):62-72. doi: 10.1093/bja/87.1.62. No abstract available. PMID 11460814
- [Background] Carr DB, Goudas LC. Acute pain. Lancet. 1999 Jun 12;353(9169):2051-8. doi: 10.1016/S0140-6736(99)03313-9. PMID 10376632
- [Background] Mulita F, Parchas N, Solou K, Tchabashvili L, Gatomati F, Iliopoulos F, Maroulis I. Postoperative Pain Scores After Open Inguinal Hernia Repair: Comparison of Three Postoperative Analgesic Regimens. Med Arch. 2020 Oct;74(5):355-358. doi: 10.5455/medarh.2020.74.355-358. PMID 33424089
- [Background] Burton, V. and P. A.J., Comparison of open and laparoscopic inguinal hernia repair. Mini-invasive Surgery, 2021. 5(26).
- [Background] Fitzgibbons RJ Jr, Ramanan B, Arya S, Turner SA, Li X, Gibbs JO, Reda DJ; Investigators of the Original Trial. Long-term results of a randomized controlled trial of a nonoperative strategy (watchful waiting) for men with minimally symptomatic inguinal hernias. Ann Surg. 2013 Sep;258(3):508-15. doi: 10.1097/SLA.0b013e3182a19725. PMID 24022443
- [Background] Hammoud, M. and J. Gerken, Inguinal Hernia, in StatPearls. 2022: Treasure Island (FL).